CLINICAL TRIAL: NCT03036527
Title: Effects of Activity Dependent Plasticity on Recovery of Bladder and Sexual Function After Human Spinal Cord Injury
Brief Title: Recovery of Bladder and Sexual Function After Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Susan Harkema PhD, Professor and Associate Director, Kentucky Spinal Cord Injury Research Center, University of Louisville Owsley B. Frazier Chair in Neurological Rehabilitation Research Director, Frazier Rehab Institute Director of the NeuroRecovery Network, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 14.0062 Bladder Sex Fxn; 5R01HD080205 (NIH)
Record Dates: First submitted 2017-01-09; First posted 2017-01-30 (Estimated); Results first posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries
Keywords: Bladder; Sexual Function
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Activity-based locomotor training (Experimental): To understand the effects of weight-bearing activity-based locomotor therapy on bladder function and sexual function. Activity-based locomotor training interventions include locomotor step training with a harness and body-weight support, 5 days a week for a total of 80, 1-hour sessions.
  Interventions: Procedure: Activity-based locomotor training
- Activity-based stand training (Experimental): To understand the effects of weight-bearing activity-based stand therapy on bladder and sexual function. Activity-based stand training interventions include stand training with a harness and body-weight support or stand training over ground, 5 days a week for a total of 80, 1-hour sessions.
  Interventions: Procedure: Activity-based stand training
- Activity-based upper arm ergometry (Experimental): To understand the effects of non-weight-bearing activity-based stand therapy on bladder and sexual function. Activity-based upper arm ergometry interventions may include arm crank training (upper arm ergometry) in while seated in the wheelchair 5 days a week for a total of 80, 1-hour sessions.
  Interventions: Procedure: Activity-based upper arm ergometry
- Activity based training + spinal epidural stimulation (Experimental): combination effect of both locomotor training and/or stand training with epidural stimulation targeting locomotion and/or stand.
  Interventions: Procedure: Activity-based locomotor training; Procedure: Activity-based stand training; Procedure: Activity-based training + spinal epidural stimulation

INTERVENTIONS:
Procedure: Activity-based locomotor training — The weight-bearing activity-based intervention will be provided via a standardized locomotor training program that is provided clinically at Frazier Rehab Institute within the NeuroRecovery Network (NRN); or similar interventions in a research protocol of stepping (IRB 07.0066).
  Other Names: Locomotor training
  Arms: Activity based training + spinal epidural stimulation; Activity-based locomotor training
Procedure: Activity-based stand training — The weight-bearing activity-based intervention will be provided via a standardized locomotor training program that is provided clinically at Frazier Rehab Institute within the NeuroRecovery Network (NRN); or similar interventions in a research protocol of stand only program (07.0268). The stand only intervention may also be provided as part of this study.
  Other Names: Stand training
  Arms: Activity based training + spinal epidural stimulation; Activity-based stand training
Procedure: Activity-based upper arm ergometry — The non-weight bearing activity-based upper arm ergometry intervention will be provided via a standardized arm crank therapy provided within this study.
  Other Names: Arm Crank
  Arms: Activity-based upper arm ergometry
Procedure: Activity-based training + spinal epidural stimulation — combination effect of both locomotor training and/or stand training with epidural stimulation targeting locomotion and/or stand.
  Arms: Activity based training + spinal epidural stimulation

SUMMARY:
Bladder and sexual dysfunction consistently ranks as one of the top disorders affecting quality of life after spinal cord injury. The insights of how activity-based training affects bladder function may prove to be useful to other patient populations with bladder and sexual dysfunction such as multiple sclerosis, Parkinson's, and stroke, as well as stimulate investigations of training's effects within other systems such as bowel dysfunction. Locomotor training could help promote functional recovery and any insights gained from these studies will enhance further investigation of the effect of bladder functioning after spinal cord injury. In addition, as suggested by a study of one of our initial participants, a reduction in the use and/or dosage of medication to enhance sexual function is a possible outcome, medications which carry risks and side effects.

DETAILED DESCRIPTION:
Objectives: To determine the effects of weight-bearing task-specific training for locomotion (stepping on a treadmill) after traumatic incomplete and complete spinal cord injury in humans on a) urodynamic parameters and b) sexual function outcomes. Weight-bearing (stand-only) and non-weight-bearing exercise (i.e. arm crank) will serve as controls.

ELIGIBILITY:
Criteria: Inclusion Criteria:

* stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate locomotor training, stand, or non-weight bearing training
* no painful musculoskeletal dysfunction,
* unhealed fracture, contracture, pressure sore or urinary tract infection that might interfere with training
* no clinically significant depression or ongoing drug abuse;
* clear indications that the period of spinal shock is concluded determined by presence of muscle tone, deep tendon reflexes or muscle spasms and discharged from standard inpatient rehabilitation
* non- progressive suprasacral spinal cord injury
* bladder and sexual dysfunction as a result of spinal cord injury

Exclusion criteria:

* unstable medical condition with cardiopulmonary disease or dysautonomia that would contraindicate locomotor training, stand, or non-weight bearing training;
* painful musculoskeletal dysfunction, unhealed fractures, contractures, pressure sores or urinary tract infections that might interfere with training
* clinically significant depression or ongoing drug abuse;
* clear indications that the period of spinal shock has not concluded and not discharged from standard inpatient rehabilitation
* progressive spinal cord injury
* no bladder and sexual dysfunction as a result of spinal cord injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Nitkin, PhD, Study Director — National Institutes of Health (NIH)
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hubscher CH, Wyles J, Gallahar A, Johnson K, Willhite A, Harkema SJ, Herrity AN. Effect of Different Forms of Activity-Based Recovery Training on Bladder, Bowel, and Sexual Function After Spinal Cord Injury. Arch Phys Med Rehabil. 2021 May;102(5):865-873. doi: 10.1016/j.apmr.2020.11.002. Epub 2020 Dec 3. PMID 33278365
- [Derived] Hubscher CH, Herrity AN, Williams CS, Montgomery LR, Willhite AM, Angeli CA, Harkema SJ. Improvements in bladder, bowel and sexual outcomes following task-specific locomotor training in human spinal cord injury. PLoS One. 2018 Jan 31;13(1):e0190998. doi: 10.1371/journal.pone.0190998. eCollection 2018. PMID 29385166

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training + Spinal Epidural Stimulation
Started | 8 | 12 | 10 | 10
Completed | 8 | 12 | 10 | 10
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Activity-based Training + Spinal Epidural Stimulation: To understand the combination effect of both locomotor training and/or stand training with epidural stimulation targeting locomotion and/or stand.
- Total: Total of all reporting groups
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training + Spinal Epidural Stimulation | Total
Number analyzed (Participants) | 8 | 12 | 10 | 10 | 40
Age, Continuous [Mean (Full Range); unit: years] | 27.4 [19 to 39] | 33.75 [19 to 50] | 31.3 [19 to 62] | 28.6 [22 to 35] | 30.8 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 2 | 7
  Male | 5 | 11 | 9 | 8 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 2
  Not Hispanic or Latino | 8 | 12 | 10 | 8 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 2 | 2 | 2 | 4 | 10
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 6 | 10 | 8 | 3 | 27
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 10 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Bladder Storage
Description: Bladder capacity (mlH2O)
Time Frame: 5 years, 2 months
Measure: Mean (Standard Deviation); unit: mLH2O
Groups:
- Activity-based Training With Spinal Epidural Stimulation: To understand the combination effect of both locomotor training and/or stand training with epidural stimulation targeting locomotion and/or stand.
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training With Spinal Epidural Stimulation
Number analyzed (Participants) | 8 | 12 | 10 | 10
mLH2O | 278.5 (147.8) | 447.75 (278.9) | 580.5 (313.2) | 313.0 (166)

2. Primary Outcome: Bladder Emptying
Description: Voiding Efficiency (% voided)
Time Frame: 5 years, 2 months
Measure: Mean (Standard Deviation); unit: % Void Efficiency
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training With Spinal Epidural Stimulation
Number analyzed (Participants) | 8 | 12 | 10 | 10
% Void Efficiency | 63.9 (8.9) | 6.2 (13.0) | 12.8 (19.8) | 28.0 (33.0)

3. Primary Outcome: Bladder Pressure
Description: Leak point pressure (cmH2O)
Time Frame: 5 years, 2 months
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training + Spinal Epidural Stimulation
Number analyzed (Participants) | 8 | 12 | 10 | 10
cm H2O | 42.7 (18.6) | 33.75 (22.7) | 45 (36.2) | 29.0 (20.0)

4. Primary Outcome: Compliance
Description: Bladder Compliance (ml/cmH2O)
Time Frame: 5 years, 2 months
Measure: Mean (Standard Deviation); unit: mL/cmH2O
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity-based Training + Spinal Epidural Stimulation
Number analyzed (Participants) | 8 | 12 | 10 | 10
mL/cmH2O | 15.5 (16.8) | 33.8 (12.5) | 17.0 (5.8) | 20.0 (25.0)

5. Secondary Outcome: International Index of Erectile Function (IIEF)
Description: There are 5 domains to the International Index of Erectile Function questionnaire: erectile function, intercourse satisfaction, orgasmic function, sexual desire, and overall satisfaction.
  Scoring 1-7: severe erectile dysfunction (ED), 8-11: Moderate ED, 12-16: mild-moderate ED, 17-21 mild ED, 22-25: no ED. Higher values represent better outcomes.
  Overall IIEF score range is 5-75; total >61.8 considered normal.
Time Frame: 5 years, 2 months
Population: Male data only (insufficient N for females)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity Based Training + Spinal Epidural Stimulation
Number analyzed (Participants) | 5 | 11 | 9 | 8
score on a scale | 20.8 (4.3) | 26.4 (5.7) | 30.0 (8.8) | 29.7 (7.6)

ADVERSE EVENTS:
Time Frame: 5 years, 2 months
Arm/Group | Activity-based Locomotor Training | Activity-based Stand Training | Activity-based Upper Arm Ergometry | Activity Based Training + Spinal Epidural Stimulation.
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/12 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/8 | 0/12 | 1/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activity-based Locomotor Training (N=8) | Activity-based Stand Training (N=12) | Activity-based Upper Arm Ergometry (N=10) | Activity Based Training + Spinal Epidural Stimulation. (N=10)
Fever (General disorders) | 0 | 0 | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Activity-based Locomotor Training (N=8) | Activity-based Stand Training (N=12) | Activity-based Upper Arm Ergometry (N=10) | Activity Based Training + Spinal Epidural Stimulation. (N=10)
Left Hand Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-09): https://cdn.clinicaltrials.gov/large-docs/27/NCT03036527/Prot_SAP_000.pdf